CLINICAL TRIAL: NCT05320900
Title: Data Construction Project for Artificial Intelligence Learning: Chest Auscultation Sound Data
Acronym: AI-sound
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Hyuk-Jae Chang, Principal Investigator, Yonsei University
Other Study IDs: AI-sound
Record Dates: First submitted 2022-03-25; First posted 2022-04-11 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Auscultation for Clinical Evaluation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Severance hospital: Cardiovascular disease patients
  Interventions: Diagnostic Test: Chest auscultation
- Yongin Severance hospital: Cardiovascular disease patients
  Interventions: Diagnostic Test: Chest auscultation
- Soon Chun Hyang University Hospital Bucheon: Cardiovascular disease patients
  Interventions: Diagnostic Test: Chest auscultation

INTERVENTIONS:
Diagnostic Test: Chest auscultation — Chest auscultation data

SUMMARY:
The purpose is to establish chest auscultation data and related clinical data for diagnosing heart and lung diseases.

DETAILED DESCRIPTION:
The incidence of cardiovascular diseases worldwide is steadily increasing. According to the report of the American Heart Association, there were 271 million cardiovascular diseases in 1990, and 523 million cases in 2019, about doubling in 30 years. The number of deaths due to cardiovascular disease is also steadily increasing from 12.1 million in 1990 to 18.6 million in 2019.

Physical examination, which is the most basic skill in patient care, consists of inspection, auscultation, percussion, and palpation. Among them, auscultation is the most widely used test in all areas where a stethoscope is used, and it is a basic examination that is essential from primary medical institutions to tertiary medical institutions for non-invasive initial diagnosis in patients complaining of chest symptoms.

However, if a specialist in the field with a lot of experience does not interpret it carefully, it is difficult to make a decision, and the deviation of the test results is large, so a significant number of patients depend on expensive follow-up tests (ultrasound, CT, MRI, etc.) This leads to a vicious cycle of incurring costs and unnecessary treatment.

Recently, with the development of machine learning techniques, computing technologies, and artificial intelligence (AI) based on a lot of data, various learning technologies are applied as tools for disease diagnosis and prognosis prediction in medicine.

Through machine learning-based chest auscultation sound analysis, there is an expectation that disease diagnosis and prognosis prediction will be able to overcome differences and interpretations by examiners. It can be very helpful in preventing overuse of tests and reducing medical costs.

ELIGIBILITY:
Inclusion Criteria:

* Adults who are 20 years and older

Exclusion Criteria:

* Patient refusal
* Uncertain radiographs
* Uncertain tests results

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who obtained chest auscultation will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Incidence of valvular heart disease | Within one week of echocardiography
  Echocardiography, coronary CTA, coronary angiography and other examinations find direct evidence of coronary artery stenosis, which can confirm the diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Hyuk-Jae Chang, MD, PhD, Principal Investigator — Severance Hospital, Yonsei University College of Medicine
Locations (3):
- South Korea (3):
  - Yongin Severance Hospital, Yŏngin, Giheung-gu
  - Soonchunhyang University Bucheon Hospital, Bucheon-si
  - Severance Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No